CLINICAL TRIAL: NCT05811286
Title: The Use of a Morcellator in Operative Hysteroscopy for Benign Intracavitary Lesions: a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S64797
Record Dates: First submitted 2023-02-07; First posted 2023-04-13 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-02

CONDITIONS: Endometrial Polyp Benign; Retained Products of Conception; Myoma;Uterus
Keywords: Endometrial polyp; Hysteroscopic surgery; Morcellation; Retained products of conception; Myoma
MeSH Terms: conditions — Myofibroma; Myoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hysteroscopic morcellation 19 Fr. intrauterine BIGATTI Shaver for uterine intracavitary lesions (Experimental): Single experimental arm of patients with a intracavitary lesion and elligible for hysteroscopic morcellation.
  Interventions: Procedure: Hysteroscopic morcellation 19 Fr. intrauterine BIGATTI Shaver for uterine intracavitary lesions

INTERVENTIONS:
Procedure: Hysteroscopic morcellation 19 Fr. intrauterine BIGATTI Shaver for uterine intracavitary lesions — With the shaver, the lesion is removed in the OR. We will include endometrial polyps, FIGO 0-1 myomas and retained products of conception.
  We will assess the completeness of hysteroscopic resection, operation time, need for cervical dilation, adverse events, pain, operator satisfaction; quality of tissue for histological examination, postoperative complications and pain.

SUMMARY:
Polyps, intracavitary myomas and retained products of conception (RPOC) are common benign intracavitary lesions of the uterus and frequently cause abnormal uterine bleeding or pain. In general, intracavitary lesions are treated by operative hysteroscopy with bipolar resectoscopic removal under general anaesthesia, performed in the theatre (OR). Potential problems with this approach are thermal damage and impairment of visibility due to loose tissue fragments necessitating multiple entries for tissue removal.

Recently, lesion morcellation by hysteroscopy has been introduced as an alternative technique. Compared to the resectoscopic approach, morcellation is reportedly associated with a shorter total procedure time, smaller fluid deficit and number of insertions. A few trials also registered a higher success rate in completeness of resection.

No significant differences in odds of surgical complications have been reported.

Most hysteroscopic morcellators have diameters up to 8 mm, for which cervical dilation under general anaesthesia is usually needed.

Recently, companies have developed hysteroscopic morcellators with smaller diameters, e.g. 6.3 mm for the 19 Fr. intrauterine BIGATTI Shaver (IBS®). This means less need for cervical dilation, and potential use without anesthesia.

At this moment, there are no prospective studies available on feasibility of the 19 Fr. intrauterine BIGATTI Shaver (IBS®). Before implementing hysteroscopic morcellation in our department, we need a feasibility study assessing the method in standard conditions in the operation room or in ambulatory setting under sedation.

Trial objectives:

Assessment of the feasibility of hysteroscopic morcellation of benign uterine intracavitary lesions. The primary objective is to assess the completeness of hysteroscopic resection in patients undergoing the procedure under general anesthesia or sedation.

Secondary objectives are to assess perioperative parameters as operation time, need for cervical dilation, adverse events, pain, operator satisfaction; to assess quality of tissue for histological examination; to assess postoperative complications and pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients:

  * Female

Ultrasonographic diagnosis of an intracavitary lesion, according the IETA terms and definitions

* endometrial polyp
* FIGO 0-1 myoma (maximum diameter 2 cm)
* RPOC (maximum diameter 2 cm, no enhanced myometrial vascularity)

Exclusion Criteria:

* • Active vaginal bleeding

  * (possible) malignancy
  * < 18y
  * Patient refusal
  * Pregnancy
  * Impossibility to access the uterine cavity (e.g. severe cervical stenosis)
  * Absence of intracavitary lesion (endometrial polyp, FIGO 0-1 myoma or RPOC) at hysteroscopy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Completeness of resection of intracavitary lesions in 50 patients, when using a hysteroscopic Bigatti Shaver. | During surgery
  If all tissue could be removed by the 19 Fr. intrauterine BIGATTI Shaver by direct visualisation at the end of the hysteroscopic procedure and at post-operative ultrasound evaluation.

SECONDARY OUTCOMES:
Operation time | During surgery
  total operation time and time necessary for the morcellation
Need for cervical dilation during procedure | During surgery
  Was it necessary to perform any dilatation with
Volume of distension fluid used / loss (deficit) during procedure | During surgery
  Deficit in fluid used during surgery?
Operator satisfaction, assessed by verbal rating scale | At the end of the procedure
  Operator satisfaction in terms of technique, ergonomics and general proceedings.
  The verbal rating scale includes Very negative; Negative; Intermediate; Positive; Very positive.
Complications | 6 weeks after surgery
  Adverse events during procedure/hospitalization and within the first 6 weeks after procedure
Pain on the first postoperative day, assessed by verbal rating scale | Day 1 post-operatively
  Pain on the first day post-operatively. The verbal rating scale includes Very negative; Negative; Intermediate; Positive; Very positive.
Histology of the intracavitary lesion | 6 weeks post-operatively
  Incidence of histological outcomes such as endometrial polyps, intracavitary myomas or remnant products of conception.
  This is a categorical variable.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Ziekenhuis Oost-Limburg, Genk
  - University Hospitals Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No
We will share general descriptive characteristics of our cohort. This includes patient and operative characteristics, final histology and patient and doctor reported outcomes.

REFERENCES:
- [Background] Munro MG, Christianson LA. Complications of Hysteroscopic and Uterine Resectoscopic Surgery. Clin Obstet Gynecol. 2015 Dec;58(4):765-97. doi: 10.1097/GRF.0000000000000146. PMID 26457853
- [Background] Shazly SA, Laughlin-Tommaso SK, Breitkopf DM, Hopkins MR, Burnett TL, Green IC, Farrell AM, Murad MH, Famuyide AO. Hysteroscopic Morcellation Versus Resection for the Treatment of Uterine Cavitary Lesions: A Systematic Review and Meta-analysis. J Minim Invasive Gynecol. 2016 Sep-Oct;23(6):867-77. doi: 10.1016/j.jmig.2016.04.013. Epub 2016 May 7. PMID 27164165
- [Background] Lee MM, Matsuzono T. Hysteroscopic intrauterine morcellation of submucosal fibroids: preliminary results in Hong Kong and comparisons with conventional hysteroscopic monopolar loop resection. Hong Kong Med J. 2016 Feb;22(1):56-61. doi: 10.12809/hkmj154600. Epub 2016 Jan 8. PMID 26744122
- [Background] Haber K, Hawkins E, Levie M, Chudnoff S. Hysteroscopic morcellation: review of the manufacturer and user facility device experience (MAUDE) database. J Minim Invasive Gynecol. 2015 Jan;22(1):110-4. doi: 10.1016/j.jmig.2014.08.008. Epub 2014 Aug 14. PMID 25128851
- [Background] Thubert T, Foulot H, Vinchant M, Santulli P, Marzouk P, Borghese B, Chapron C. Surgical treatment: Myomectomy and hysterectomy; Endoscopy: A major advancement. Best Pract Res Clin Obstet Gynaecol. 2016 Jul;34:104-21. doi: 10.1016/j.bpobgyn.2015.11.021. Epub 2016 Jun 22. PMID 27400649
- [Background] Pakrashi T. New hysteroscopic techniques for submucosal uterine fibroids. Curr Opin Obstet Gynecol. 2014 Aug;26(4):308-13. doi: 10.1097/GCO.0000000000000076. PMID 24950124
- [Background] Vidal-Mazo C, Forero-Diaz C, Lopez-Gonzalez E, Yera-Gilabert M, Machancoses FH. Clinical recurrence of submucosal myoma after a mechanical hysteroscopic myomectomy: Review after 5 years follow up. Eur J Obstet Gynecol Reprod Biol. 2019 Dec;243:41-45. doi: 10.1016/j.ejogrb.2019.10.014. Epub 2019 Oct 21. PMID 31671290
- [Background] van Dongen H, Emanuel MH, Wolterbeek R, Trimbos JB, Jansen FW. Hysteroscopic morcellator for removal of intrauterine polyps and myomas: a randomized controlled pilot study among residents in training. J Minim Invasive Gynecol. 2008 Jul-Aug;15(4):466-71. doi: 10.1016/j.jmig.2008.02.002. Epub 2008 Apr 18. PMID 18588849
- [Background] AlHilli MM, Nixon KE, Hopkins MR, Weaver AL, Laughlin-Tommaso SK, Famuyide AO. Long-term outcomes after intrauterine morcellation vs hysteroscopic resection of endometrial polyps. J Minim Invasive Gynecol. 2013 Mar-Apr;20(2):215-21. doi: 10.1016/j.jmig.2012.10.013. Epub 2013 Jan 5. PMID 23295201
- [Background] Li C, Dai Z, Gong Y, Xie B, Wang B. A systematic review and meta-analysis of randomized controlled trials comparing hysteroscopic morcellation with resectoscopy for patients with endometrial lesions. Int J Gynaecol Obstet. 2017 Jan;136(1):6-12. doi: 10.1002/ijgo.12012. Epub 2016 Nov 7. PMID 28099700
- [Background] Stoll F, Lecointre L, Meyer N, Faller E, Host A, Hummel M, Boisrame T, Akladios C, Garbin O. Randomized Study Comparing a Reusable Morcellator with a Resectoscope in the Hysteroscopic Treatment of Uterine Polyps: The RESMO Study. J Minim Invasive Gynecol. 2021 Apr;28(4):801-810. doi: 10.1016/j.jmig.2020.07.007. Epub 2020 Jul 16. PMID 32681995
- [Background] Ansari SH, Bigatti G, Aghssa MM. Operative hysteroscopy with the Bigatti shaver (IBS (R)) for the removal of placental remnants. Facts Views Vis Obgyn. 2018 Sep;10(3):153-159. PMID 31191850
- [Background] Bigatti G, Ansari SH, Di W. The 19 Fr. Intrauterine Bigatti Shaver (IBS(R)): a clinical and technical update. Facts Views Vis Obgyn. 2018 Sep;10(3):161-164. PMID 31191851